CLINICAL TRIAL: NCT03955263
Title: Prevalence of Asymptomatic Malaria During Pregnancy and Its Effect on Pregnancy Outcomes in Women Attending Antenatal Clinic in Central India
Brief Title: Malaria In Pregnancy in Central India
Acronym: MIP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Lata Medical Research Foundation, Nagpur (Other)
Responsible Party: Sponsor
Other Study IDs: RPC#30
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Pregnant Women
Keywords: asymptomatic; Malaria; pregnancy; prevalence; RT-PCR
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Dried Blood Spots
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present study is planned to be conducted at a district level women and children's hospital at Nagpur with the following objectives:

Objectives:

i) To assess the prevalence of asymptomatic malaria infection with all four species of malarial parasites namely P. falciparum, P. malariae, P. ovale and P. vivax during the first/second trimester of pregnancy among women attending the antenatal clinic at a secondary level urban health facility using PCR (polymerase chain reaction) for malaria parasites.

ii) To determine the effect of malaria on duration of pregnancy, adverse outcomes and birth outcomes at delivery

DETAILED DESCRIPTION:
Public Health Rationale:

Despite comprehensive malaria control programmes, control measures specifically aimed at malaria in pregnancy are not adequately available. The epidemiological data are scanty in order to develop effective policies to address this problem. The major barrier to successful eradication or elimination of malaria transmission is the inability to detect and treat asymptomatic carriers of the malarial parasites. Asymptomatic carriers do not seek treatment for infection and thus the life cycle of the infection continues. The systematic identification and treatment of individuals with asymptomatic P.falciparum and P. vivax, as part of a surveillance intervention strategy, are important for reducing the parasite reservoir and would help to decrease transmission of the disease. Data on asymptomatic carriage is not available from India.

Routine screening for malaria and anaemia followed by prompt management should be encouraged to curb the effect of malaria and anaemia on the pregnant women as well as her fetus. The present study is planned to be conducted at a district level women and children's hospital at Nagpur with the following objectives:

Objectives:

i) To assess the prevalence of asymptomatic malaria infection with all four species of malarial parasites namely P. falciparum, P. malariae, P. ovale and P. vivax during the first/second trimester of pregnancy among women attending the antenatal clinic at a secondary level urban health facility using PCR (polymerase chain reaction) for malaria parasites.

ii) To determine the effect of malaria on duration of pregnancy, adverse outcomes and birth outcomes at delivery

Study Design And Study Population:

This is a prospective cohort study of pregnant women in their first/second trimester of pregnancy attending the antenatal clinic at a secondary level healthcare facility at Nagpur, India.

Investigators propose collecting a two-three dried blood spot (DBS) sample for all enrolled women and symptomatic (fever with or without chills) neonates and infants at enrollment when the haemoglobin measurement is performed. Asymptomatic parasitaemia will be detected using a dual-antigen rapid diagnostic kit (RDK), microscopy, and species-specific PCR. PCR for the detection of malaria parasite would be performed at the National Institute for Research in Tribal Health (NIRTH) at Jabalpur, India

ELIGIBILITY:
Inclusion Criteria:

- Pregnant woman in first / second trimester of pregnancy

Exclusion Criteria:

* Pregnant woman in first / second trimester of pregnancy those do not consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women in their first / second trimester attending Antenatal clinics at district level women and children's hospital at Nagpur
Sampling Method: Probability Sample
Enrollment: 887 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Asymptomatic parasitaemia | January 2019 to December 2019
  Number of women having asymptomatic malaria which will be detected using a dual-antigen rapid diagnostic kit (RDK), microscopy, and species-specific PCR. PCR for the detection of malaria parasite would be performed at the National Institute for Research in Tribal Health (NIRTH) at Jabalpur, India.
Effect of malaria on duration of pregnancy | January 2019 to December 2019
  Difference in mean gestational age at delivery or end of pregnancy among women with versus those without RT-PCR-confirmed malaria infection during pregnancy.
Outcome of the pregnancy | January 2019 to December 2019
  Number of live births, still birth / miscarriage, elective termination / death after delivery
Birth weight | January 2019 to December 2019
  Difference in mean birth weight among all infants and among term singleton infants born to women with versus those without RT-PCR-confirmed malaria infection during pregnancy
Infant Outcome | January 2019 to December 2019
  Number of episode of Fever till 42 days of infant age among all infants and among term singleton infants born to women with versus those without RT-PCR-confirmed malaria infection during pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Archana Patel, MD, PhD, Principal Investigator — Program Director and CFO, Lata Medical Research Foundation
Locations (1):
- Lata Medical Research Foundation, Nagpur, Maharashtra, India